CLINICAL TRIAL: NCT02760004
Title: PRogram In Support of Moms: An Innovative Stepped-Care Approach for Obstetrics and Gynecology Clinics
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Byatt, Associate Professor of Psychiatry and Obstetrics & Gynecology, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H00009163; 1U01DP006093 (NIH)
Record Dates: First submitted 2016-04-27; First posted 2016-05-03 (Estimated); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prism Intervention (Experimental): PRogram In Support of Moms (PRISM)
  Interventions: Behavioral: PRogram In Support of Moms (PRISM)
- MCPAP for Moms Intervention (Experimental): MCPAP for Moms (Massachusetts Child Psychiatry Access Program for Moms)
  Interventions: Behavioral: MCPAP for Moms

INTERVENTIONS:
Behavioral: PRogram In Support of Moms (PRISM) — * Access to MCPAP for Moms
  * PRogram In Support of Moms Toolkit with Stepped Care Algorithms
  * Support clinic specific implementation using the Addressing Problems Through Organizational Change (APTOC) platform
  * Customization of depression screening for each practice
  * Proactively engage and track all women who screen +ve on the Edinburgh Postnatal Depression Scale(EPDS)
  * Employ psychoeducation and Motivational Interviewing to engage patients with depression
  * medical assistant champion and psychiatrist contact bi-weekly to review cases
  * Stepped care treatment to depression screening/assessment
  Other Names: Rapid Access to Perinatal Psychiatric care in Depression
  Arms: Prism Intervention
Behavioral: MCPAP for Moms — * 30-60 minute presentation on perinatal depression
  * Access to telephonic psychiatric consultation with MCPAP for Moms perinatal psychiatrist for Ob/Gyns
  * Access to Ob/Gyn provider assessment and treatment recommendations via one-time face-face MCPAP for Moms psychiatrist patient evaluation
  * Access to assessment and treatment protocols in Provider Toolkit
  * Resource provision/referrals
  Arms: MCPAP for Moms Intervention

SUMMARY:
The primary goal of this study is to develop, evaluate, and share a new low-cost program for Obstetrics/Gynecology (Ob/Gyn) practices which will help to improve depression treatment for women during pregnancy and after childbirth.

DETAILED DESCRIPTION:
Upwards of 1 in 5 women suffer from depression during pregnancy or within a year after giving birth. It has negative effects on birth outcomes, infant attachment, and children's behavior/development. Maternal suicide causes 20% of postpartum deaths in depressed women. Although the vast majority of perinatal women are amenable to being screened for depression, screening alone does not improve treatment rates or patient outcomes. Ob/Gyn practices need supports in place to adequately address depression in their patient populations. Thus, the Investigators developed and pilot tested the PRogram In Support of Moms (PRISM), to create a comprehensive intervention that is proactive, multifaceted, and practical. PRISM aims to improve perinatal depression treatment and treatment response rates through: (1) access to immediate resource provision/referrals and psychiatric telephone consultation for Ob/Gyn providers; (2) clinic-specific implementation of stepped care, including training support and toolkits; and, (3) proactive treatment engagement, patient monitoring, and stepped treatment response to depression screening/assessment. PRISM builds on a low-cost and widely disseminated population-based model for delivering psychiatric care in primary care settings developed by our team. Because it uses existing infrastructure and resources, PRISM, has the potential to be feasible, sustainable, and transportable to other practice settings. The Investigators will compare PRISM vs. MCPAP for Moms which provides access to resource provision/referrals and psychiatric telephone consultation, in a clinical trial in which Investigators will randomize 10 Ob/Gyn practices to either PRISM or MCPAP for Moms (Massachusetts Child Psychiatry Access Program for Moms) - intervention. Patient participants will participate in either PRISM or MCPAP for Moms, depending on what intervention their practice is assigned to. The Investigators will compare the effectiveness of PRISM vs. MCPAP for Moms to improve depression severity and treatment participation in pregnancy through 13 months postpartum among 340 patients (n=170/group).

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18-55 years
3. English speaking
4. >4 weeks Gestational age (GA) until 4 months postpartum
5. Receiving care from one of the 10 participating practices (five will participate in PRISM (intervention group) and five will have access to MCPAP For Moms (comparison group)
6. Edinburgh Postnatal Depression Scale score (EPDS) ≥10
7. Able to communicate in written and spoken English; and
8. Cognitively able to participate in informed verbal consent

Exclusion Criteria:

1. Lack of verbal and written English fluency
2. Under age 18 or over age 55
3. substance use disorder as determined by the questions in 4 Ps questionnaire
4. Screen positive for bipolar disorder via the Mood Disorder Questionnaire (MDQ)
5. Prisoner
6. Women participating in 'Moms do care' study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 312 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Byatt, DO, MS, MBA, Principal Investigator — University of Massachusetts Medical School/UMass Memorial Health Care; Tiffany A Moore Simas, MD, MPH, MEd, Principal Investigator — University of Massachusetts Medical School/UMass Memorial Health Care; Jeroan J Allison, MD, MS, Principal Investigator — University of Massachusetts Medical School/UMass Memorial Health Care
Locations (1):
- UMass Medical School/UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing plan is as applicable with CDC requirements and policy. All IPD that underlie results in a publication will be shared. Analysis of the data by approved researchers will only be conducted as delineated in the approved proposal. Only the minimum amount of data necessary to accomplish the proposed analysis will be released and must be destroyed after the specified analysis has been completed. All analyses will be subjected to independent verification.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after main publication up to a period of 3 years.
Access Criteria: All researchers who work with the PRISM data will submit a proposal and sign a data-sharing agreement. Researchers will first submit a proposal which will be reviewed by the PRISM Publication Committee. If the proposal is approved, the researcher will sign a data-sharing agreement in which they commit to 1) using the data only for research purposes, 2) keeping the data secure using proper technological precautions, 3) destroying the data after analyses are completed, and 4) only conduct analyses described in the approved proposal.
  Our research team will create de-identified analytical datasets and share them with approved researchers as .CSV files that will be transferred by secure encrypted transfer using a secure managed data transfer server.

REFERENCES:
- [Background] Hirschfeld RM, Williams JB, Spitzer RL, Calabrese JR, Flynn L, Keck PE Jr, Lewis L, McElroy SL, Post RM, Rapport DJ, Russell JM, Sachs GS, Zajecka J. Development and validation of a screening instrument for bipolar spectrum disorder: the Mood Disorder Questionnaire. Am J Psychiatry. 2000 Nov;157(11):1873-5. doi: 10.1176/appi.ajp.157.11.1873. PMID 11058490
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Chen H, Wang J, Ch'ng YC, Mingoo R, Lee T, Ong J. Identifying mothers with postpartum depression early: integrating perinatal mental health care into the obstetric setting. ISRN Obstet Gynecol. 2011;2011:309189. doi: 10.5402/2011/309189. Epub 2011 Sep 15. PMID 21941662
- [Background] Flynn HA, O'Mahen HA, Massey L, Marcus S. The impact of a brief obstetrics clinic-based intervention on treatment use for perinatal depression. J Womens Health (Larchmt). 2006 Dec;15(10):1195-204. doi: 10.1089/jwh.2006.15.1195. PMID 17199460
- [Background] Burton A, Patel S, Kaminsky L, Rosario GD, Young R, Fitzsimmons A, Canterino JC. Depression in pregnancy: time of screening and access to psychiatric care. J Matern Fetal Neonatal Med. 2011 Nov;24(11):1321-4. doi: 10.3109/14767058.2010.547234. Epub 2011 Jan 24. PMID 21261444
- [Background] Goodman JH, Tyer-Viola L. Detection, treatment, and referral of perinatal depression and anxiety by obstetrical providers. J Womens Health (Larchmt). 2010 Mar;19(3):477-90. doi: 10.1089/jwh.2008.1352. PMID 20156110
- [Background] Glavin K, Smith L, Sorum R, Ellefsen B. Redesigned community postpartum care to prevent and treat postpartum depression in women--a one-year follow-up study. J Clin Nurs. 2010 Nov;19(21-22):3051-62. doi: 10.1111/j.1365-2702.2010.03332.x. Epub 2010 Aug 19. PMID 20726926
- [Background] Glavin K, Smith L, Sorum R. Prevalence of postpartum depression in two municipalities in Norway. Scand J Caring Sci. 2009 Dec;23(4):705-10. doi: 10.1111/j.1471-6712.2008.00667.x. Epub 2009 Aug 29. PMID 19490523
- [Background] Chaudron LH, Kitzman HJ, Peifer KL, Morrow S, Perez LM, Newman MC. Prevalence of maternal depressive symptoms in low-income Hispanic women. J Clin Psychiatry. 2005 Apr;66(4):418-23. doi: 10.4088/jcp.v66n0402. PMID 15816782
- [Background] Delucchi KL, Tajima B, Guydish J. Development of the Smoking Knowledge, Attitudes, and Practices (S-KAP) Instrument. J Drug Issues. 2009 Mar;39(2):347-364. doi: 10.1177/002204260903900207. PMID 20717496
- [Background] McDonald SD, Calhoun PS. The diagnostic accuracy of the PTSD checklist: a critical review. Clin Psychol Rev. 2010 Dec;30(8):976-87. doi: 10.1016/j.cpr.2010.06.012. Epub 2010 Jul 6. PMID 20705376
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Swanson LM, Flynn HA, Wilburn K, Marcus S, Armitage R. Maternal mood and sleep in children of women at risk for perinatal depression. Arch Womens Ment Health. 2010 Dec;13(6):531-4. doi: 10.1007/s00737-010-0177-z. Epub 2010 Jul 14. PMID 20628772
- [Background] Clement S, Brohan E, Jeffery D, Henderson C, Hatch SL, Thornicroft G. Development and psychometric properties the Barriers to Access to Care Evaluation scale (BACE) related to people with mental ill health. BMC Psychiatry. 2012 Jun 20;12:36. doi: 10.1186/1471-244X-12-36. PMID 22546012
- [Background] Cooper LA, Brown C, Vu HT, Palenchar DR, Gonzales JJ, Ford DE, Powe NR. Primary care patients' opinions regarding the importance of various aspects of care for depression. Gen Hosp Psychiatry. 2000 May-Jun;22(3):163-73. doi: 10.1016/s0163-8343(00)00073-6. PMID 10880709
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Heitjan DF. Annotation: what can be done about missing data? Approaches to imputation. Am J Public Health. 1997 Apr;87(4):548-50. doi: 10.2105/ajph.87.4.548. No abstract available. PMID 9146428
- [Background] Myers ER, Aubuchon-Endsley N, Bastian LA, Gierisch JM, Kemper AR, Swamy GK, Wald MF, McBroom AJ, Lallinger KR, Gray RN, Green C, Sanders GD. Efficacy and Safety of Screening for Postpartum Depression [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Apr. Report No.: 13-EHC064-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK137724/ PMID 23678510
- [Background] Weathers F, Litz B, Huska J, Keane T. PTSD checklist-civilian version. In. Boston: Nation Center for PTSD. Behavioral Sciences Division. ; 1994
- [Background] Little R. Statistical Analysis with Missing Data. New York: John Wiley and Sons; 1987
- [Background] Karlson K, Holm A. Decomposing primary and secondary effects: A new decomposition method. Research in Social Stratification and Mobility 2011;29:221-37.
- [Derived] Julce C, Flahive J, Lightbourne T, Podila S, Mahanna A, Zimmermann M, Sheldrick RC, Moore Simas TA, Byatt N. Descriptive Characteristics of Psychiatric Medication Discontinuation Among Perinatal Women With Depressive Symptoms. Early Interv Psychiatry. 2025 Jun;19(6):e70070. doi: 10.1111/eip.70070. PMID 40539750
- [Derived] Byatt N, Brenckle L, Sankaran P, Flahive J, Ko JY, Robbins CL, Zimmermann M, Allison J, Person S, Moore Simas TA. Effectiveness of two systems-level interventions to address perinatal depression in obstetric settings (PRISM): an active-controlled cluster-randomised trial. Lancet Public Health. 2024 Jan;9(1):e35-e46. doi: 10.1016/S2468-2667(23)00268-2. PMID 38176840
- [Derived] Schipani Bailey E, Byatt N, Carroll S, Brenckle L, Sankaran P, Kroll-Desrosiers A, Smith NA, Allison J, Simas TAM. Results of a Statewide Survey of Obstetric Clinician Depression Practices. J Womens Health (Larchmt). 2022 May;31(5):675-681. doi: 10.1089/jwh.2021.0147. Epub 2021 Sep 2. PMID 34491103
- [Derived] Masters GA, Brenckle L, Sankaran P, Person SD, Allison J, Moore Simas TA, Ko JY, Robbins CL, Marsh W, Byatt N. Positive screening rates for bipolar disorder in pregnant and postpartum women and associated risk factors. Gen Hosp Psychiatry. 2019 Nov-Dec;61:53-59. doi: 10.1016/j.genhosppsych.2019.09.002. Epub 2019 Oct 22. PMID 31710859
- [Derived] Moore Simas TA, Brenckle L, Sankaran P, Masters GA, Person S, Weinreb L, Ko JY, Robbins CL, Allison J, Byatt N. The PRogram In Support of Moms (PRISM): study protocol for a cluster randomized controlled trial of two active interventions addressing perinatal depression in obstetric settings. BMC Pregnancy Childbirth. 2019 Jul 22;19(1):256. doi: 10.1186/s12884-019-2387-3. PMID 31331292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from the 10 participating OB/Gyn practices from October 2017 to November 2020. The 10 obstetric practices were randomized to one of the two interventions (5 each) and patient participants from these practices provided data for evaluating the effectiveness of each intervention. Individual patient participant data were analyzed to assess effectiveness.
Pre-assignment Details: Of the 1265 screened, 312 met the inclusion criteria. The practices were randomized to the 2 intervention arms of the study.
Units Other Than Participants: OB Practices
Groups:
- PRISM Intervention: PRogram In Support of Moms (PRISM)
  PRogram In Support of Moms (PRISM): • Access to MCPAP for Moms
  * PRogram In Support of Moms Toolkit with Stepped Care Algorithms
  * Support clinic specific implementation using the Addressing Problems Through Organizational Change (APTOC) platform
  * Customization of depression screening for each practice
  * Proactively engage and track all women who screen +ve on the Edinburgh Postnatal Depression Scale(EPDS)
  * Employ psychoeducation and Motivational Interviewing to engage patients with depression
  * medical assistant champion and psychiatrist contact bi-weekly to review cases
  * Stepped care treatment to depression screening/assessment
- MCPAP for Moms: MCPAP for Moms
  Access to MCPAP for Moms: • 30-60 minute presentation on perinatal depression
  * Access to telephonic psychiatric consultation with MCPAP for Moms perinatal psychiatrist for Ob/Gyns
  * Access to Ob/Gyn provider assessment and treatment recommendations via one-time face-face MCPAP for Moms psychiatrist patient evaluation
  * Access to assessment and treatment protocols in Provider Toolkit
  * Resource provision/referrals
Period: Overall Study
Arm/Group | PRISM Intervention | MCPAP for Moms
Started | 150; 5 OB Practices | 162; 5 OB Practices
Completed | 137; 5 OB Practices | 140; 5 OB Practices
Not Completed | 13; 0 OB Practices | 22; 0 OB Practices
Not completed — Lost to Follow-up | 13 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRISM Intervention | MCPAP for Moms | Total
Number analyzed (Participants) | 150 | 162 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6) | 33 (6) | 32 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 162 | 312
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 47 | 91
  Not Hispanic or Latino | 104 | 115 | 219
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 4 | 16 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 26 | 13 | 39
  White | 82 | 102 | 184
  More than one race | 12 | 15 | 27
  Unknown or Not Reported | 22 | 15 | 37
Region of Enrollment [Number; unit: participants]
  United States | 150 | 162 | 312
Education [Count of Participants; unit: Participants]
  Grade school/Some high school | 9 | 6 | 15
  High school diplomaor GED equivalent | 46 | 32 | 78
  Some college no degree | 34 | 43 | 77
  Associate degree | 8 | 15 | 23
  Bachelor's degree | 30 | 21 | 51
  Master's degree | 22 | 29 | 51
  Doctoral degree or equivalent | 0 | 15 | 15
  Other - Missing data | 1 | 1 | 2
Primary source of payment for prenatal care [Count of Participants; unit: Participants]
  Tricare/Self-pay/Other | 2 | 2 | 4
  Private or Commercial | 61 | 82 | 143
  Medicaid/Mass Health/Other public | 86 | 78 | 164
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Edinburgh Postnatal Depression Scale Score (EPDS)
Description: EPDS - Edinburgh Postnatal Depression Scale is an instrument used to measure depression. The score range is 0 to 30. A higher score means more depressed. Depressed perinatal patients receiving care from practices enrolled in PRISM will experience more improvement in depression symptoms than patients receiving care from the MCPAP for Moms practices (2 point difference-of-difference in EPDS).
Time Frame: Baseline up to 13 months postpartum
Population: Out of the participants enrolled in the study, data was obtained and analyzed for 118 participants in the PRISM Intervention and 117 in the MCPAP for Moms for this outcome measure. These subgroups are based on the number of Participants who had both the baseline EPDS score and a final 11-13 months postpartum EPDS score. Participants can enter at [0 -20 weeks GA, 20-40 weeks GA or 0-12 weeks postpartum] and this serves as Baseline. Final measurement occurs at 11 to 13 months postpartum.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PRISM Intervention: PRogram In Support of Moms (PRISM)
  PRogram In Support of Moms (PRISM): • PRogram In Support of Moms Toolkit with Stepped Care Algorithms
  * Support clinic specific implementation using the Addressing Problems Through Organizational Change (APTOC) platform
  * Customization of depression screening for each practice
  * Proactively engage and track all women who screen +ve on the Edinburgh Postnatal Depression Scale(EPDS)
  * Employ psychoeducation and Motivational Interviewing to engage patients with depression
  * medical assistant champion and psychiatrist contact bi-weekly to review cases
  * Stepped care treatment to depression screening/assessment
- MCPAP for Moms: MCPAP for Moms
  * 30-60 minute presentation on perinatal depression
  * Access to telephonic psychiatric consultation with MCPAP for Moms perinatal psychiatrist for Ob/Gyns
  * Access to Ob/Gyn provider assessment and treatment recommendations via one-time face-face MCPAP for Moms psychiatrist patient evaluation
  * Access to assessment and treatment protocols in Provider Toolkit
  * Resource provision/referrals
Arm/Group | PRISM Intervention | MCPAP for Moms
Number analyzed (Participants) | 118 | 117
score on a scale | -4.3 (4.5) | -4.2 (5.2)

2. Secondary Outcome: Participants Initiating Treatment
Description: Number of depressed perinatal patients receiving care from practices enrolled in PRISM who initiated treatment measured by attendance (i,e. one initial mental health assessment or treatment visit) as compared to women receiving care from practices enrolled in MCPAP for Moms.
Time Frame: Baseline to up to 13 months postpartum
Population: Participants can enter at [0 -20 weeks GA, 20-40 weeks GA or 0-12 weeks postpartum] and this serves as Baseline. Final measurement occurs at 11 to 13 months postpartum.
Measure: Count of Participants; unit: Participants
Arm/Group | PRISM Intervention | MCPAP for Moms
Number analyzed (Participants) | 150 | 162
Participants | 78 | 70

3. Secondary Outcome: Participants Sustaining Mental Health Treatment
Description: Sustainment of mental health treatment for depressed perinatal patients receiving care from practices enrolled in PRISM. as measured an average ≥1 mental health visit every 1 month until remission of symptoms or study assessment) as compared to women receiving care from practices enrolled in MCPAP for Moms.
Time Frame: Baseline to up to 13 months postpartum
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PRISM Intervention | MCPAP for Moms
Number analyzed (Participants) | 150 | 162
Participants | 38 | 32

ADVERSE EVENTS:
Time Frame: 37 months - throughout the enrollment period
Arm/Group | PRISM Intervention | MCPAP for Moms
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/162
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/162
Other Adverse Events (participants affected / at risk) | 0/150 | 1/162
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRISM Intervention (N=150) | MCPAP for Moms (N=162)
Hospitalization for suicidal risk (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT02760004/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT02760004/SAP_001.pdf